CLINICAL TRIAL: NCT06523634
Title: Salvage Stereotactic Body Radiotherapy of the Prostate Bed for Biochemical Recurrence After Radical Prostatectomy.
Acronym: STEREOBED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE3764
Record Dates: First submitted 2024-05-28; First posted 2024-07-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard of care radiotherapy
  Interventions: Radiation: SOC RT
- SBRT (Experimental): SBRT: 5 fractions
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — 5 fractions of SBRT to the prostate bed with or without whole pelvic radiotherapy Treatment every other day.
  Arms: SBRT
Radiation: SOC RT — Standard salvage radiotherapy to the prostate bed with or without whole pelvic radiotherapy. Each participating centre can specify upfront which RT schedule will be used in the control arm, with the choice between the following schedules:
  * Hypofractionated: 20 fractions (Daily treatment (OTT 4-5 weeks))
  * Normofractionated: 32-35 fractions (Daily treatment (OTT 7-8 weeks))
  Arms: Control

SUMMARY:
This is a a randomized phase II/III trial comparing salvage SBRT with standard of care (SOC) regimens for patients with a persistent detectable PSA or biochemical progression during follow-up after radical prostatectomy.

DETAILED DESCRIPTION:
This is a multicentric randomized seamless phase II/III study comparing SBRT to conventional RT or moderately hypofractionated RT on the prostate bed.

All subjects will be randomly assigned in a 1:1 ratio:

1. Experimental arm: Radiotherapy treatment in 5 fractions.
2. Control arm: Radiotherapy treatment within a normofractionated or mildly hypofractionated schedule. For the control arm, each participating center can choose between a normofractionated schedule (32 to 35 treatment sessions) and a moderately hypofractionated schedule (20 sessions).

ELIGIBILITY:
INCLUSION CRITERIA

1. Localized adenocarcinoma (cN0M0) of the prostate treated primarily with radical prostatectomy with definitive intent.
2. Either persistent PSA after prostatectomy (PSA ≥ 0.1 ng/mL at least 6 weeks after prostatectomy), or biochemical progression (two consecutive rising PSA amounts with a PSA >0.1 ng/mL , or three consecutive PSA rises)
3. WHO PS 0-1
4. Age ≥18 years
5. Ability to understand and willingness to sign a study-specific informed consent prior to study entry
6. Ability to understand and answer the EPIC-26 form in one of the languages available

EXCLUSION CRITERIA

1. Patients with a pT4 tumor at prostatectomy
2. Patients with previously pathologically confirmed N1
3. Patients with macroscopically involved margin at surgery (R2)
4. Patients with a history of distant metastases
5. Patients with a recurrence visible on imaging (local, pelvic, or distant). Pelvic nodes with a small diameter >1cm and/or positive on PSMA without other explanation, are considered as a pelvic recurrence.
6. Latest PSA > 2ng/ml
7. Patients with a IPSS >20
8. Gleason 10 tumor
9. Prior history of high-intensity focused ultrasound ablation (HIFU), cryosurgery or brachytherapy of the prostate
10. Prior pelvic radiotherapy
11. Prior hormonal therapy started more than 6 weeks before randomization
12. History of inflammatory bowel disease, ataxia telangiectasia, prior rectal or bladder surgery.
13. Other active malignancy, except non-melanoma skin cancer, superficial bladder cancer, or malignancies with a documented disease-free survival for a minimum of 3 years before randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
SBRT impact on patient-reported GI and GU symptoms | 2 years post treatment
  Urinary and bowel domain of the EPIC-26 (Expanded Prostate Cancer Index Composite).

SECONDARY OUTCOMES:
Patient Reported Outcomes | at end of RT and following time-points counted from start of RT : 4-7 weeks (only in experimental arm), 3 months, 6 months, 1 year and yearly up to 5 years
  Patient-reported outcomes according to the different
  * EPIC-26 domains (0-100)
  * IPSS score (0-35)
  * EQ-5D-5L scores (five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression)
Ccost-utility during radiotherapy | during radiotherapy
  Cost-utility analysis based on EQ-5D-5L (five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression)versus costs of RT and transportation during radiotherapy
Physician-scored toxicity | up to 5 years
  Physician-scored toxicity according to CTCAE 5.0 (grades) (Early: within 90 days; or late: 90 or more days after SBRT). Proportion of patients with G2+ toxicity will be reported specifically.
Blood lymphocyte evolution between study arms | 5 years
  Lymphocyte count nadir relative to baseline
To compare biochemical progression-free survival (bPFS) to historical control and between study arms | 5 years
  Biochemical progression-free survival (bPFS)
To compare local and regional recurrences between study arms, up to 5 years. | 5 years
  Local and regional control
To compare Overall survival (OS) between study arms, up to 5 years. | 5 years
  Overall survival (OS)
To compare distant metastases-free survival (dmFS) between study arms | 5 years
  Distant metastases-free survival (dmFS).

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (12):
  - AZorg, Aalst
  - GZA Ziekenhuis ZAS Kempenstraat, Antwerp
  - Ziekenhuis Aan de Stroom (ZAS), Antwerp
  - AZ Sint Jan, Bruges
  - Jules Bordet Institute, H.U.B, Brussels
  - Ziekenhuis Oost-Limburg (ZOL) Campus Sint-Jan, Genk
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - CHU HELORA - Hôpital de La Louvière - site Jolimont, La Louvière
  - AZ Sint-Maarten, Mechelen
  - CHU UCL Namur - Site Elisabeth, Namur
  - Cliniques universitaires Saint-Luc (UCLouvain), Woluwe-Saint-Lambert

IPD SHARING:
Plan to Share IPD: No